CLINICAL TRIAL: NCT05758337
Title: Clinical and Functional Rationalization of the Use of Vibropneumostimulation in the Rehabilitation System of Patients After Dental Implantation
Brief Title: Vibropneumostimulation in the Rehabilitation After Dental Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 190
Record Dates: First submitted 2023-02-08; First posted 2023-03-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-09

CONDITIONS: Dental Implantation
Keywords: dental implantation; vibropneumostimulation

STUDY DESIGN:
Intervention Model Description: The first group is a group of subjects on whom, after implantation, a new technique was applied, including the effect of vibropneumostimulation on the pereimplant tissues
Who Masked: Participant
Masking Description: The second is a group of subjects whose rehabilitation was carried out by the well-known classical method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group with exposure of vibropneumostimulation (Experimental): The first group is a group of subjects on whom, after implantation, a new technique was applied, including the effect of vibropneumostimulation on the pereimplant tissues.
  Interventions: Device: Vibropneumostimulation
- A group of standart therapy (No Intervention): The second is a group of subjects whose rehabilitation was carried out by the well-known classical method.

INTERVENTIONS:
Device: Vibropneumostimulation — New vibrators and techniques of vibropneumostimulation of periimplant tissues have been developed, which will allow us to develop a new concept of the relationship of bone remodulation processes around implants of various designs.
  Arms: A group with exposure of vibropneumostimulation

SUMMARY:
A new comprehensive technique of dental implantation and rehabilitation of patients will be developed and theoretically justified, including an individual dental implant of a dowel system made of non-woven titanium material with through porosity and vibropneumostimulation, which will improve the functional and anatomical results of treatment.

In the complex treatment and rehabilitation of patients after dental implantation, a vibropneumostimulator with vibratodes of its own design will be used, which activate bone remodeling, which will expand the practical application and theoretical knowledge in the field of hardware massage.

DETAILED DESCRIPTION:
The aim of the study: to improve the results of treatment of patients after dental implantation by using vibropneumostimulation of periimplant tissues.

In the work, a complex of functional and clinical methods (thermography, radiography, periotestometry) will be used. The following methods will also be used:

* echosteometry, thanks to which the density of bone tissue in the periimplant zone will be studied, which will allow to study the processes of bone tissue remodulation.
* radioisotope diagnostics, thanks to which the dynamics of bone metabolism processes around implants will be studied, which will expand the knowledge of the metabolism of jaw bones.

The subject of the study is the remodulation of bone tissue around the implant, which will allow us to develop a new concept of the relationship of processes in the bone tissue around implants of various designs. The study is based on the study and generalization of existing scientific data on surgical treatment of patients, as well as on the assessment of the relevance and degree of development of the topic. To improve the quality of care for patients after implantation, in our research we will use vibro-pneumatic action on the tissues of the upper and lower jaws in the field of implantation by a device of the SamSMU design - a medical vibro-pneumatic stimulator, it will be an automated system for pneumatic wave massage and vibration exposure.

A vibropneumostimulator with vibratodes of its own design will be introduced into clinical practice, which will expand the arsenal of hardware treatment of an implantologist.

In the complex treatment of patients with partial and complete loss of teeth, an improved dental implant of a dowel system made of non-woven titanium material with through porosity will be offered for using.

ELIGIBILITY:
Inclusion Criteria:

* patients with a history of previous unsuccessful implantations,
* patients with a history of bad habits,
* patients with low bone density (CT),
* patients who have sinus lifting surgery performed simultaneously

Exclusion Criteria: No

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
restoration of dentition by installing crowns on the installed implants | 4 months
  implant stability according to the method of Resonance Frequency Analysis that register magnetic vibrations of the pin together with the implant in the form of an indicator Implant Stability Quotient

SECONDARY OUTCOMES:
installation of the gumformer | 7 months
  rate of patients with installation of the gumformer on the installed implants according to the X-ray
the beginning of the functional load | 7 months
  rate of patients with the beginning of the functional load on the restored dentition according to the X-ray

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Bayrikov, MD, Study Director — Samara State Medical University
Locations (1):
- Samara state medical university, Samara, Russia